CLINICAL TRIAL: NCT05237726
Title: Comparison of the Efficacy and Safety for Different Regimen of Venous Thromboembolism Pharmacoprophylaxis Among Severely Burn Patients
Brief Title: Efficacy and Safety for Different Regimen of VTE Pharmacoprophylaxis Among Severely Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, KHALID ALSULAIMAN, Dr. Khalid Al Sulaiman, Consultant, Critical Care Clinical Pharmacist, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC18-400-R
Record Dates: First submitted 2022-01-03; First posted 2022-02-14 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Burns
Keywords: Severely burn; BSA≥20%; Enoxaparin; Unfractionated Heparin; VTE; Bleeding
MeSH Terms: conditions — Burns; Hemorrhage | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Intervention Model Description: Three groups randomized to receive DVT prophylaxis either enoxaparin 30 mg every 12 hours, enoxaparin 40 mg once daily and unfractionated heparin 5000 units every 8 hours
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Unfractionated Heparin (UFH) 5000 U q8 hours (Active Comparator): Severely burn injuries (BSA≥20%) will receive Unfractionated Heparin (UFH) 5000 U q8 hours as pharmacological VTE prophylaxis
  Interventions: Drug: Unfractionated heparin 5000 U q8 hours
- Enoxaparin 40 mg q24 hours (Active Comparator): Severely burn injuries (BSA≥20%) will receive Enoxaparin 40 mg q24 hours as pharmacological VTE prophylaxis
  Interventions: Drug: Enoxaparin 40 mg q24 hours
- Enoxaparin 30 mg q12 hours (Active Comparator): Severely burn injuries (BSA≥20%) will receive Enoxaparin 30 mg q12 hours as pharmacological VTE prophylaxis
  Interventions: Drug: Enoxaparin 30 mg q12 hours

INTERVENTIONS:
Drug: Enoxaparin 40 mg q24 hours — Severely burn injuries (BSA≥20%) will be assigned to 3 modality regimens of pharmacological VTE prophylaxis: Unfractionated heparin 5000 U SQ q8 hours, Enoxaparin 40 mg SQ q24 hours or Enoxaparin 30 mg SQ q12 hours.
  Arms: Enoxaparin 40 mg q24 hours
Drug: Enoxaparin 30 mg q12 hours — Severely burn injuries (BSA≥20%) will be assigned to 3 modality regimens of pharmacological VTE prophylaxis: Unfractionated heparin 5000 U SQ q8 hours, Enoxaparin 40 mg SQ q24 hours or Enoxaparin 30 mg SQ q12 hours.
  Arms: Enoxaparin 30 mg q12 hours
Drug: Unfractionated heparin 5000 U q8 hours — Severely burn injuries (BSA≥20%) will be assigned to 3 modality regimens of pharmacological VTE prophylaxis: Unfractionated heparin 5000 U SQ q8 hours, Enoxaparin 40 mg SQ q24 hours or Enoxaparin 30 mg SQ q12 hours.
  Arms: Unfractionated Heparin (UFH) 5000 U q8 hours

SUMMARY:
This study aims to assess the feasibility and safety of VTE prophylaxis for 3 modality regimens (Unfractionated heparin 5000 U SQ q8 hours, Enoxaparin 40 mg SQ q24 hours or Enoxaparin 30 mg SQ q12 hours) in adult patients (≥18 y/o) with severely burn injuries (BSA≥20%) by measuring the bleeding incidence and VTE events.

DETAILED DESCRIPTION:
This is a pilot , randomized control trial-Open label, prospective trial in tertiary academic hospitals for patient admitted to burn ICU for at least 24 hours of injury or transferred from other hospital(s) within 7 days of injury. Each patient admitted meets the inclusion criteria will be randomize by block randomization to either receive heparin 5000 units S.C. TID, enoxaparin 40 mg S.C. OD, or Enoxaparin 30 mg S.C. BID. VTE prophylaxis should be started within 36 hours of injury, if the patient is transferred from another facility, VTE prophylaxis should be started immediately unless contraindicated. All patients should undergo diagnostic ultrasound at baseline ( before starting the prophylaxis) to assess any presence of DVT and as clinically indicated for clinical suspicion for VTE thereafter until discharge, an urgent spiral CTA chest will be requested on clinical suspicion for PE. Anti Xa factor will be monitored at day 3, and weekly thereafter until discharge unless there is active bleeding or high clinical suspicion for bleeding. Will follow-up patient until discharge from ICU, developed VTE requiring treatment (switch to treatment dose), developed HIT or death.

ELIGIBILITY:
Inclusion Criteria:

* Burn ICU admitted adult patients, age ≥ 18 years old.
* Body Mass Index of 18.5 to < 40 kg/m2.
* TBSA of 20% or more.

Exclusion Criteria:

* VTE history.
* Death within 24 hours of injury.
* Burn injuries combined with trauma requiring withholding pharmacoprophylaxis more than 48 hours.
* Coagulopathy (INR > 1.7, PTT> 2 times upper normal limit, platelet < 50k mm3)
* Patient with positive baseline US for VTE.
* Heparin induced thrombocytopenia (HIT).
* Active bleeding.
* Patients with CrCl of 30 ml/min or less.
* Patients using anticoagulation treatment dose for other indications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding events (major and minor) | Through study completion, an average of 2 years
  Daily assessment of major and minor Bleeding. Bleeding will classified into major and minor bleeding. Major bleeding defined as clinically overt bleeding associated with a fall ≥Hb 20g/L, transfusion of ≥2U PRBC or whole blood, retroperitoneal or intracranial bleeding or requiring urgent medical intervention. Minor bleeding defined as those not fulfilling the criteria of major or clinically significant bleeding.
Adverse effects in surgical outcomes (i.e. Graft loss, donor site morbidity, requirement of hemostatic intervention). | Through study completion, an average of 2 years
  Daily assessment of donor site and graft site bleeding/failure.
  Graft site bleeding defined as bleeding at skin graft recipient site that requires premature wound exploration ( before 3 days postoperatively), bed side or operating room intervention to stop bleeding ( stitching, hemostatic agent or cauterization) with or without blood transfusion.
  Donor site bleeding/hematoma is any bleeding leading to a drop in hemoglobin > 2 grams, hemodynamic instability or bleeding requiring urgent transfusion.
  Graft failure due to hematoma that require re-grafting or more than 50% of the graft site.
  Enoxaparin should be held 12 hours and unfractionated heparin 3-4 hours before percutaneous tracheostomy OR epidural catheter if indicated.
Recruitment and consent rates | Through study completion, an average of 2 years
  To assess the recruitment and consent rate to evaluate trial feasibility

SECONDARY OUTCOMES:
Target anti Xa factor for enoxaparin or unfractionated heparin in severely burn patients. | Through study completion, an average of 2 years
  Anti-Xa: Blood samples for Anti-Xa were obtained day 3 after patient is admitted to ICU (Plasma sample will be collected in blue tube "no citrate" ~ 5 mL/Test), then Anti-Xa obtained weekly thereafter until discharge. Anti-Xa obtained immediately 4 hours after administration of Enoxaparin and 3 hours after administration of unfractionated Heparin
Incidence of Heparin induced thrombocytopenia (HIT). | Through study completion, an average of 2 years
Number of days that patients stay in hospital | Through study completion, an average of 2 years
  The length of an inpatient episode of care, calculated from the day of admission in hospital to day of discharge/death
Number of patients died within intensive care unit stay | Through study completion, an average of 2 years
  The number of deaths of patients admitted to the intensive care unit (ICU), divided by the number of patient discharges from the ICU (including deaths and transfers).
Incidence of VTE events (Symptomatic) | Through study completion, an average of 2 years
  All patients participating in the study should undergo bilateral lower extremity duplex scan to rule out DVT at baseline before starting VTE prophylaxis and as clinically indicated for clinical suspicion for VTE thereafter until discharge from ICU, developing VTE incident or death.
  Urgent spiral CTA chest will be requested on clinical suspicion for PE.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Sulaiman KA, Al-Ramahi G, Aljuhani O, Al-Joudi K, Alhujayri AK, Al-Shomer F, Silas J, Al Dabbagh T, Al Harbi S, AlDekhayel S, Eldali A, Alqahtani R, Vishwakarma R, Al-Dorzi HM. Comparison of the safety and efficacy for different regimens of pharmaco-prophylaxis among severely burned patients: a randomized controlled trial. Eur J Trauma Emerg Surg. 2024 Apr;50(2):567-579. doi: 10.1007/s00068-024-02443-9. Epub 2024 Jan 19. PMID 38240791